CLINICAL TRIAL: NCT00050297
Title: YM598 in Patients With Rising PSA After Initial Therapy for Localized Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Astellas Pharma US, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 598-CL-004
Record Dates: First submitted 2002-12-03; First posted 2002-12-04 (Estimated); Last update posted 2012-06-07 (Estimated); Status verified 2012-06

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — N-(6-methoxy-5-(2-methoxyphenoxy)-2-(pyrimidin-2-yl)pyrimidin-4-yl)-2-phenylethenesulfonamide

INTERVENTIONS:
Drug: YM598

SUMMARY:
The purpose of this study is to determine the optimal dosage of YM598 for slowing down disease progression in patients with rising PSA after initial therapy for localized prostate cancer.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Study Completion 2004-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (23):
- Belgium (2):
  - University Clinic AZ, Brussels
  - University Clinic UCL St. Luc, Brussels
- Czechia (4):
  - Private Urology Out-patient Ward, Jablonec nad Nisou
  - Clinic of Urology, University Hospital, Králové
  - Clinic of Urology, University Hospital, Olomouc
  - Clinic of Urology, University Hospital, Prague
- Hôpital Bichat, service de Urology, Paris, France
- Germany (4):
  - Haingasse 22, Bad Homburg
  - Klinik und Poliklinik für Urologie, Universitätsklinikum Carl-Gustav-Carus, Dresden
  - Klinik u. Poliklinik für Urologie, Philipps Universität, Baldingerstraße, Marburg
  - Krummbogen 15, Marburg
- Poland (5):
  - Regional Hospital, Department of Urology, Bydgoszcz
  - MedSource Poland, Gdansk
  - Bielanski Hospital, Department of Urology, Warsaw
  - Oncology Center, Department of Urinary Tract Cancer, Warsaw
  - Medical University, Clinic of Urology, Wroclaw
- Spain (3):
  - Complejo Hospitaliaro Juan Canalejo, Servicio de Urología, Corunna
  - Fundacion Hospital Alcorcón, Servicio Urología, Madrid
  - Hospital Universitario Principe de Asturias, Servicio de Urología, Ctra., Madrid
- United Kingdom (4):
  - Department of Urology, Bristol Royal Infirmary, Bristol
  - Department of Urology, Gartnavel Hospital, Glasgow
  - Department of Urology, Norfolk & Norwich Hospital, Norwich
  - Department of Urology, Taunton & Somerset Hospital, Taunton